CLINICAL TRIAL: NCT01796314
Title: Impact of a Therapeutic Educational Programme for Alzheimer's Disease Patients and Their Caregiver in Community Dwelling, on the AD Patient's Quality of Life
Brief Title: Impact of Therapeutic Educational Programme on the Alzheimer's Disease Affected Patient's Quality of Life
Acronym: THERAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC31/11/255; PREQHOS n°11 255 07 (Other Grant/Funding Number: Ministry of Health)
Record Dates: First submitted 2013-02-19; First posted 2013-02-21 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Alzheimer Disease
Keywords: Therapeutic educational programme for Alzheimer's disease patients and their caregiver; Alzheimer's disease, mild to moderately severe stages; Community dwelling patients with family caregiver; quality of life
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A : intervention (Experimental): 85 dyads "patient/caregiver" in witch the patient suffers from mild to moderately severe Alzheimer's disease patients (MMSE 11 to 26), and lives at home with a caregiver
  Interventions: Behavioral: Therapeutic Educational Program
- Group B : Control (No Intervention): There si no associated intervention

INTERVENTIONS:
Behavioral: Therapeutic Educational Program — The intervention is a therapeutic educational programme as recommended in the care of Alzheimer's disease. It includes two consultations for the dyad AD patient/caregiver and four group sessions, one a week, for caregivers only. The intervention length is 2 months.
  These collective sessions focus on :
  1. Knowledge of the disease
  2. Pharmacological and non pharmacological treatments. Behavioural and psychological symptoms of dementia
  3. Crisis situations. Prevention of caregiver's exhaustion
  4. Assistive devices and care pathways.
  Monitoring will consist of a two consultations to 6 and 12 months including assessment of secondary outcome measures.
  Other Names: Therapeutic education programme
  Arms: Group A : intervention

SUMMARY:
Therapeutic education expands in Alzheimer's Disease management in France. Several studies revealed a positive impact on caregiver's burden and/or quality of life. The purpose of this study, is to determine whether a therapeutic educational programme for both AD patients and primary caregivers, in community dwelling, improves patient's quality of life.

DETAILED DESCRIPTION:
This study is designed to determine whether a therapeutic educational programme for both AD patients, in community dwelling, and their primary caregivers improves patient's quality of life, after two months.

Design : This study is a monocentric randomised controlled intervention trial

Population : One hundred and seventy dyads 'patient-caregiver' in which the patient suffers from mild to moderately severe Alzheimer's disease patients (MMSE 11 to 26), lives in community dwelling and has a primary caregiver will be included during eighteen months. The primary caregiver is define as a person living with the patient or providing care at least 3 times a week or 8 hours per week; he/she isn't a professional. Eighty five dyad will be include in the intervention group (group A) and eighty five in the control group (group B).

Outcome : Our primary endpoint is the AD patient's quality of life assessed by Logsdon's Quality of life in Alzheimer's Disease scale (Qol-AD) reported by the caregiver at two months.

Our secondary endpoints are caregiver's burden assessed by the Zarit Burden Inventory, frequency and severity of behavioural and psychological symptoms assessed by the Neuro Psychiatric Inventory, independence in personal and instrumental daily life activities assessed by Katz's Activities of Daily Living and Lawton's Instrumental Activities of Daily Living scales, and caregiver's quality of life assessed by the Nottingham Health Profile at 6 months. The patient quality of life will also be recorded at 12 months on the logsdon's Quality of Life in Alzheimer's Disease scale reported, and at every visit (MO, M2, M6, et M12) on the same scale dut (QoL-AD) reported by the patient himself.

Intervention :

The intervention is a therapeutic educational programme. It includes two consultations for the dyad AD patient/caregiver and four group sessions, one a week, for caregivers only. The intervention length is 2 months.

The intervention group (n=85) will benefit from an educational programme that includes two consultations for the dyad AD patient/caregiver and four group sessions for caregivers only. The two consultations will be held at baseline (MO) and two months later (M2); the first one (MO)will include : the 'educational diagnosis', the comprehensive assessment of the patient and assessment of the judgement criteria. Between MO and M2 the primary caregivers will participate to four collective sessions one per week about, of 3 hours length : 1- Knowledge of the disease; 2- Pharmacological and non pharmacological treatments. Behavioural and psychological symptoms of dementia 3- Crisis situations. Prevention of caregiver's exhaustion 4- Assistive devices and care pathways. At M2, the dyad will benefit from : assessment of response to the educational objectives and of the judgement criteria.

The control group (n=85) will benefit from routine care.

The intervention will be implemented over an eighteen month period.

Monitoring will consist of a two consultations to 6 and 12 months including assessment of primary and secondary judgment criteria.

Data collection :

Data will be collected in Access data basis and SAS software will be used to perform statistic analysis. Intention to treat analysis using linear mixed model will be performed, adjusting for patient (disease severity), caregiver characteristics (burden) and occurence of life event that may interfere with the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patient suffering from mild to moderately severe Alzheimer's disease patients (MMSE 11 to 26)
* in community dwelling
* with an informal caregiver (person living with the patient or providing care 3 times a week or 8 hours per week)
* is informed and has given his/her consent
* whom caregiver is informed and has given his/her consent

Exclusion Criteria:

* patient with other type of dementia
* living in nursing home or long term care
* with no caregiver
* not informed or has not given his/her consent
* whom caregiver is not informed or has not given his/her consent

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2013-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease patient's quality of life | 2 months
  Alzheimer's Disease patient's quality of life assessed by Logsdon's Quality of life in Alzheimer's Disease scale (QoL-AD) reported by the caregiver

SECONDARY OUTCOMES:
Caregiver quality of life | 2, 6 and 12 months
  * Caregiver's burden assessed by the Zarit Burden Inventory
  * Frequency and severity of behavioural and psychological symptoms assessed by the Neuro Psychiatric inventory
  * Independence in personal and instrumental daily life activities assessed by Katz's Activities of Daily Living and Lawton's Instrumental Activities of Daily Living scales
  * Caregiver's quality of life assessed by the Nottingham Health Profile at 6 months
  * Patient quality of life at 6 and 12 months on the Logsdon's Quality of Life in Alzheimer's Disease scale reported by the caregiver
  * Patient quality of life at 2,6 and 12 months on the Logsdon's Quality of Life in Alzheimer's Disease scale reported by the patient himself

CONTACTS AND LOCATIONS:
Overall Officials: Hélène VILLARS, MD, Principal Investigator
Locations (1):
- CHU de Toulouse, Hôtel-Dieu, 2 rue Viguerie, Toulouse, France

REFERENCES:
- [Result] Villars H, Cantet C, de Peretti E, Perrin A, Soto-Martin M, Gardette V. Impact of an educational programme on Alzheimer's disease patients' quality of life: results of the randomized controlled trial THERAD. Alzheimers Res Ther. 2021 Sep 12;13(1):152. doi: 10.1186/s13195-021-00896-3. PMID 34511121
- [Derived] Villars H, Gardette V, Perrin A, Hein C, Elmalem S, de Peretti E, Zueras A, Vellas B, Nourhashemi F. Study protocol: Randomised controlled trial to evaluate the impact of an educational programme on Alzheimer's disease patients' quality of life. Alzheimers Res Ther. 2014 Oct 27;6(5-8):66. doi: 10.1186/s13195-014-0066-1. eCollection 2014. PMID 25478028